CLINICAL TRIAL: NCT06415513
Title: The Effect of Autonomous Sensory Meridian Response (ASMR) Videos on Sleep Quality and Stress Levels of Nursing Students Before First Clinical Practice
Brief Title: The Effect of (ASMR) Videos on Sleep Quality and Stress Levels on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Ayşe Kabuk, Asst. Prof., Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23.02.2024/420449
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Students; Nursing
Keywords: Autonomous Sensory Meridian Response; anxiety; sleep
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: intervention group: Autonomous Sensory Meridian Response; control group: no intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): For 7 days, they were asked to watch ASMR videos for 20-30 minutes every evening at 22:00 before going to bed. The videos were downloaded to the student's computer or phone in advance, the student was asked to switch his/her phone to airplane mode to block the stimuli during the viewing, to watch these videos with headphones, to reduce the sounds in the room as much as possible, to lie on his/her bed and to wear comfortable clothes.
  Interventions: Other: ASMR
- control (No Intervention): no intervention

INTERVENTIONS:
Other: ASMR — We used 7 ASMR videos published on the most watched ASMR channel on the YouTube platform, in which applications such as hair combing, brushing, massaging the head are applied sequentially and repeatedly, and there is no speech.
  Arms: intervention

SUMMARY:
This study was planned to evaluate the effect of Autonomous Sensory Meridian Response (ASMR) videos on sleep quality and stress levels of nursing students before clinical practice.

DETAILED DESCRIPTION:
Autonomous Sensory Meridian Response (ASMR) is a physiological phenomenon that describes a tingling sensation caused by specific visual and auditory triggers, usually starting on the scalp and travelling down the body. These trigger stimuli are often socially intimate in nature and often involve repetition of movements and/or sounds.

According to studies conducted among university students, it is generally stated that university students have poor sleep quality and sleep inadequately. Negative impact on students' sleep quality is a factor that causes them to experience stress. Nursing students are faced with an important source of stress due to the various situations they encounter in the education and practice processes. Although clinical education offers rich opportunities to gain hands-on experience, it is reported that the clinical component of nursing education provides the highest source of stress for nursing students.

This study was planned to evaluate the effect of Autonomous Sensory Meridian Response (ASMR) videos on sleep quality and stress levels of nursing students before clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years,
* illiterate,
* volunteer to participate in the study
* First-year nursing students who have not done clinical practice before

Exclusion Criteria:

* have done clinical practice before

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-05-11 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
sleep quality | In the study, The sleep quality of the students in the intervention group was measured before the interventions and on the 8th day after the 7-day interventions. Sleep quality of the students in the control group was measured on day 1 and day 8.
  PUKI was accepted in determining sleep quality, and in 1989 and its validity and reliability were determined (Cronbach's alpha=0.80). In our country, the validity and reliability study was carried out by Ağargün et al. (16) and the Cronbach alpha value of the scale was found to be 0.80. The scale is a four-point Likert type and contains a total of 24 questions; subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), use of sleeping pills (component 6) and daytime dysfunction (component 3) 7) consists of 7 components. The sum of the seven component scores gives the total PUKI score. The response of each is scored between 0-3 according to symptom frequency. The total score has a value between 0-21.
anxiety | In the study, The anxiety of the students in the intervention group was measured before the interventions and on the 8th day after the 7-day interventions. Anxiety of the students in the control group was measured on day 1 and day 8.
  State - Trait Anxiety Inventory-STAI. It was developed by Spielberger et al. (1970). The scale consists of two parts: the State Anxiety Inventory and Trait Anxiety Inventory. The State Anxiety Inventory determines how the individual feels at a certain moment and under certain conditions, and the Trait Anxiety Inventory determines how the individual feels regardless of the situation and conditions. Each scale contains two types of statements with 20 items. In the state anxiety scale, the responses were evaluated with a 4-point scale (never, a little, a lot, completely). In the trait anxiety scale, the answers of the participants were measured with a 4-point scale (never, sometimes, very often, almost always). The total score value obtained from both scales varies between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayşe Kabuk, Zonguldak, Kozlu/Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ı want to share my research protocol after six months.

REFERENCES:
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Stinson C, Curl ED, Hale G, Knight S, Pipkins C, Hall I, White K, Thompson N, Wright C. Mindfulness Meditation and Anxiety in Nursing Students. Nurs Educ Perspect. 2020 Jul/Aug;41(4):244-245. doi: 10.1097/01.NEP.0000000000000635. PMID 32168090
- [Result] Smejka T, Wiggs L. The effects of Autonomous Sensory Meridian Response (ASMR) videos on arousal and mood in adults with and without depression and insomnia. J Affect Disord. 2022 Mar 15;301:60-67. doi: 10.1016/j.jad.2021.12.015. Epub 2021 Dec 13. PMID 34915083